CLINICAL TRIAL: NCT03843515
Title: "Safety and Tolerability of Neoadjuvant Nivolumab for Locally Advanced Resectable Oral Cancer Combined With [18F] BMS-986192 / [18F] -FDG PET Imaging and Immunomonitoring for Response Prediction"
Brief Title: Neoadjuvant Nivolumab for Oral Cancer Combined With FDG and Anti-PD-L1 PET/CT Imaging for Response Prediction
Acronym: NeoNivo
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, C. Menke- van der Houven van Oordt, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-002643
Record Dates: First submitted 2019-02-13; First posted 2019-02-18 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Oral Cavity Squamous Cell Carcinoma
Keywords: head and neck squamous cell carcinoma; nivolumab; PD-L1; PET/CT; neoadjuvant
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Phase I safety and feasibility study with additional pilot biomarker assessments
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant nivolumab (Experimental): All subject will receive 400mg flat dose nivolumab in the neoadjuvant setting
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Neoadjuvant nivolumab flat dose 400mg
  Other Names: Neoadjuvant nivolumab

SUMMARY:
Safety and tolerability of neoadjuvant nivolumab for locally advanced resectable oral cancer, combined with [18F]BMS-986192 / [18F]-FDG PET imaging and immunomonitoring for response prediction

DETAILED DESCRIPTION:
Intensive treatment regimens with surgical resection and adjuvant (chemo)radiotherapy of patients with locally advanced oral cancer still result in only 50-60% cure rate, leaving a substantial group of patients who will develop a local recurrence or distant metastases with minimal curative salvage treatment options. Treatment with anti-PD-1 monoclonal antibodies (mAbs) has shown promise in patients with recurrent/metastatic head and neck squamous cell carcinoma (r/m HNSCC). This supports the hypothesis that including treatment with anti PD-1 mAb nivolumab could improve the outcome for patients with locally advanced oral cancer resulting in a higher cure rate. Response rate with nivolumab was below 20% in unselected patients with r/m HNSCC. Therefore, biomarkers for response are urgently needed. Tumor PD-L1 immunohistochemistry (IHC) was shown to be related to nivolumab response but cannot be reliably used for patient selection. Temporal and spatial heterogeneity of tumor PD-L1 expression (within and between tumor lesions) might be responsible for its suboptimal predictive value as biomarker of response. Therefore there is a need to further evaluate tumor PD-L1 expression as predictive biomarker, as well as exploring alternatives. Serial PET imaging with [18F]BMS-986192 (anti-PD-L1 tracer) and [18F]-FDG has the potential to provide whole body information of the patient over time, at baseline as well as on treatment and represents a biomarker for toxicity and efficacy. In addition, we will investigate the immunophenotype of the patient and tumor, as well as the presence of neoantigens and other potential other biomarkers such as plasma vesicle miRNAs.

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically confirmed diagnosis of locally advanced oral cancer (stage III/IV) which is planned for treatment with curative intent including surgical resection.
2. Be willing and able to provide written informed consent/assent for the trial.
3. Be more then 18 years of age on day of signing informed consent.
4. Must agree to provide tissue from fresh tumor biopsy pretreatment and from the surgical resection material to determine the actual PD-L1 status and perform immunomonitoring/DNA/RNA profiling.
5. Willing to allow up to two additional biopsies when baseline [18F]BMS-986192 PET /[18F]-FDG PET scans show heterogeneous and/or discrepant uptake.
6. Have a performance status of 0-1 on the ECOG Performance Scale (Appendix 2).
7. Demonstrate adequate organ function as defined in table 1. All screening labs should be performed within 2 weeks before any study imaging procedures are performed
8. Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception during the study and for 23 weeks after the last dose of nivolumab. Women who are not of childbearing potential (i.e. who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception (Appendix 4)
9. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception during the study and for 31 weeks after the last dose of nivolumab (Appendix 4).

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent within 4 weeks of the first dose of treatment or has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
2. Has had another known invasive malignancy within the previous 5 years and/or has had surgery, chemotherapy, targeted small molecule therapy or radiation therapy within 5 years for a known malignancy prior to study day 0.
3. Has a known current additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
4. If subject received major surgery for any other reason, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
5. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of day -5. Inhaled or topical steroids, and adrenal replacement steroid > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
6. Has an active autoimmune disease requiring systemic steroid treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids.
7. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
8. Has an active infection requiring systemic therapy.
9. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
10. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
11. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 23 weeks after the last dose of trial treatment.
12. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways.
13. Has a known history of Human Immunodeficiency Virus (HIV) infection (HIV 1/2 antibodies).
14. Has known active Hepatitis B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
(Serious) adverse events | untill 100 days after last study drug administration
  Adverse events
SUV values | 2 years
  SUVpeak/mean/max of tumor lesions on FDG-PET/anti-PD-L1 PET

SECONDARY OUTCOMES:
Correlation between PET data and Blood/Tissue markers | 2 years
  The correlation between continuous values as SUV and the categorical variables tissue PD-1 and PD-L1 IHC will be assessed for each tumor lesion. Correlation with immuno-monitoring analysis in tumor tissue/lymph nodes and blood, plasma vesicle miRNAs from blood, as well as DNA/RNA profiling in tumor tissue at baseline and at surgery will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: C. W. Menke, Phd, MD, Principal Investigator — Amsterdam UMC, location VUmc; C. R. Leemans, Phd, MD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University medical center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No